CLINICAL TRIAL: NCT00027547
Title: Nonmyeloablative Allogeneic Hematopoietic Cell Transplantation From HLA Matched Sibling Donors For Treatment Of Patients With High Risk Acute Lymphocytic Leukemia In Complete Remission
Brief Title: Combination Chemotherapy and Total-Body Irradiation Followed by Peripheral Stem Cell or Bone Marrow Transplantation in Treating Patients With Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 1586.00; FHCRC-1586.00; NCI-H01-0080; CDR0000069042 (Registry Identifier: PDQ)
Record Dates: First submitted 2001-12-07; First posted 2003-01-27 (Estimated); Last update posted 2011-11-30 (Estimated); Status verified 2011-11

CONDITIONS: Leukemia
Keywords: adult acute lymphoblastic leukemia in remission; childhood acute lymphoblastic leukemia in remission
MeSH Terms: conditions — Leukemia | interventions — Cyclosporine; Cytarabine; fludarabine phosphate; Methotrexate; Mycophenolic Acid; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Biological: therapeutic allogeneic lymphocytes
Drug: cyclosporine
Drug: cytarabine
Drug: fludarabine phosphate
Drug: methotrexate
Drug: mycophenolate mofetil
Procedure: allogeneic bone marrow transplantation
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Peripheral stem cell transplantation may be able to replace immune cells that were destroyed by chemotherapy and radiation therapy. Sometimes the transplanted cells are rejected by the body's normal tissues. Mycophenolate mofetil and donor white blood cells may prevent this from happening.

PURPOSE: Phase I/II trial to determine the effectiveness of combination chemotherapy and total-body irradiation followed by peripheral stem cell transplantation in treating patients who have acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine if a one-year disease free survival of 40% and a day 200 transplant-related mortality of less than 25% can be achieved in patients with high-risk acute lymphoblastic leukemia in complete remission treated with a nonmyeloablative conditioning regimen comprising fludarabine and total body irradiation followed by allogeneic peripheral blood stem cell or bone marrow transplantation.
* Evaluate the efficacy and toxicity of donor lymphocyte infusion in the treatment of minimal residual disease after nonmyeloablative allografting in these patients.

OUTLINE: This is a multicenter study.

Patients receive a nonmyeloablative conditioning regimen comprising fludarabine IV on days -4 to -2 and total body irradiation (TBI) on day 0. Children undergo allogeneic peripheral blood stem cell transplantation (PBSCT) or bone marrow transplantation after TBI on day 0. Adults undergo filgrastim (G-CSF)-mobilized allogeneic PBSCT after TBI on day 0.

Patients also receive graft-versus-host disease (GVHD) prophylaxis therapy comprising oral cyclosporine twice daily on days -3 to 56 and then tapered and oral mycophenolate mofetil once at 5-10 hours after transplantation on day 0 and then twice daily on days 1-27.

Patients who have no evidence of grade 2 or greater acute GVHD or clinically extensive chronic GVHD, have been off GVHD prophylaxis therapy for 1-2 weeks, and have stable or increasing minimal residual disease after discontinuation of GVHD prophylaxis therapy receive donor lymphocyte infusion (DLI) IV over 30 minutes. DLI repeats every 4 weeks for a total of 3 doses (if necessary).

Patients without a history of CNS leukemia and patients with a history of CNS leukemia previously treated with prophylactic craniospinal irradiation receive methotrexate (MTX) or cytarabine (ARA-C) intrathecally (IT) for a total of 2 doses before transplantation and for a total of 6 doses beginning on day 32 after transplantation. Patients with a history of CNS leukemia not previously treated with craniospinal irradiation undergo craniospinal irradiation for 11 days before conditioning regimen and then MTX or ARA-C IT for a total of 6 doses beginning on day 32 after transplantation. Male patients also undergo testicular radiotherapy for 7 days.

Patients are followed at 1, 2, 3, 6, 12, 18, and 24 months.

PROJECTED ACCRUAL: A total of 30 patients (20 adults and 10 children) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute lymphoblastic leukemia (ALL)
* Adult patients must meet 1 of the following criteria:

  * Age 50 to 75 with high-risk ALL in complete remission (CR) (less than 5% blasts by morphology on bone marrow aspirate and absence of peripheral blasts) or ALL in second CR (CR2) or greater
  * Age 18 to 50 with high-risk ALL in first CR (CR1) and either ineligible for conventional allogeneic transplantation (based on general medical condition) or refused conventional transplantation

    * High-risk adult ALL in CR1 includes patients meeting 1 or more of the following criteria:

      * Age 30 and over
      * Non-T-cell phenotype
      * Cytogenetic abnormalities including t(9;22), t(4;11), trisomy 8, or monosomy 7
      * Failure to achieve CR after 4 weeks of induction chemotherapy
  * Age 18 to 50 with ALL in CR2 or greater and ineligible for conventional allogeneic transplantation based on general medical condition
  * Age 18 to 50 with high-risk ALL in CR2 or greater and refused conventional allogeneic transplantation
* Pediatric patients must meet 1 of the following criteria:

  * Under age 18 with high-risk ALL in CR1 and ineligible for conventional allogeneic transplantation based on general medical condition

    * High-risk pediatric ALL in CR1 includes patients meeting 1 or more of the following criteria:

      * Cytogenetic abnormalities

        * t(9;22) with WBC at least 25,000/mm3 at diagnosis
        * t(4;11) in patients under age 1 or age 10 and over
        * Hypodiploidy (no more than 45 chromosomes)
      * Failure to achieve CR after 4 weeks of induction chemotherapy
      * Persistent peripheral blasts after 1 week of induction chemotherapy
  * Under age 18 with CR2 or greater and ineligible for conventional allogeneic transplantation based on general medical condition
  * Age 12 and under allowed if approved by the principle investigator
* No active CNS disease
* Availability of a sibling donor (excluding an identical twin)

  * HLA genotypically identical for at least 1 haplotype
  * HLA-A, -B, -C, -DRB1, and -DQB1 genotypically or phenotypically identical

PATIENT CHARACTERISTICS:

Age:

* See Disease Characteristics
* 75 and under

Performance status:

* Karnofsky 50-100% (adults)
* Lansky 40-100% (children)

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics

Hepatic:

* No fulminant liver failure
* No alcoholic hepatitis
* No history of bleeding esophageal varices
* No grade II or greater hepatic encephalopathy
* No hepatic synthetic dysfunction evidenced by prolongation of PT with INR greater than 2.5
* No intractable ascites related to portal hypertension
* No bacterial or fungal liver abscess
* No chronic viral hepatitis with bilirubin greater than 5 mg/dL
* No biliary obstruction with bilirubin greater than 5 mg/dL
* No concurrent symptomatic biliary disease

Renal:

* Not specified

Cardiovascular:

* Cardiac ejection fraction at least 30%

Pulmonary:

* No requirement for supplementary continuous oxygen

Other:

* HIV negative
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 1 year after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent posttransplantation growth factors during mycophenolate mofetil administration

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-07; Study Completion 2004-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Georges, MD, Study Chair — Fred Hutchinson Cancer Center
Locations (3):
- United States (2):
  - Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Universitaet Leipzig, Leipzig, Germany